CLINICAL TRIAL: NCT00231504
Title: Study of Follicle Stimulating Hormone (FSH) Receptor in Women With Low Antral Follicle Count
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe Aucan, Department Clinical Rechearch of Developpement
Other Study IDs: P041013; CRC04140
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2007-03

CONDITIONS: Antral Follicle Deficit; Fertility
Keywords: Polymorphism P1; Polymorphism P2; FSH Receptor; Antral follicle count; FSH receptor polymorphism
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood samples — Blood samples

SUMMARY:
The deficit in the total number of antral follicles is associated with a reduction of the ovarian fertility potential in young women.

The principal objective of this study is to evaluate the relationship between FSH receptor polymorphism and antral follicle count.

The investigators have designed a study of FSH receptor polymorphisms P1 and P2 as an association with a low antral follicle count in the ovary.

DETAILED DESCRIPTION:
The present study will compare the prevalence of FSH receptor polymorphisms P1 and P2 in women having reduced follicle count (1 to 9 antral follicles) or normal follicle count (13 to 20 antral follicles) determined by ultrasound scans.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years old
* 1 to 9 or 13 to 20 antral follicles
* Caucasian, occidental Europe
* Presence of both ovaries
* Informed consent

Exclusion Criteria:

* Ovarian anomalies
* Menopause
* Pregnancy
* Other diseases

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: YOUNG WOMAN
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2005-10; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato FANCHIN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Antoine Beclere Hospital, Obstetrics and Gynaecology and Reproduction Medicine Service, Paris, France